CLINICAL TRIAL: NCT04360005
Title: Managed Access Programs for ABL001, Asciminib
Status: Available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CABL001A02401M
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Chronic Myeloid Leukemia in Chronic Phase
Keywords: Chronic myeloid leukemia; CML; CML-CP; Asciminib; ABL001
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — asciminib

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Asciminib — Patients receive Asciminib
  Other Names: ABL001

SUMMARY:
The purpose of this registration form is to list all Managed Access Programs (MAPs) related to ABL001, asciminib

ELIGIBILITY:
Inclusion Criteria:

1. An independent request was received from a licensed physician.
2. The patient has a serious or life-threatening disease or condition and there is no comparable or satisfactory alternative therapy available for diagnosis, monitoring, or treatment.
3. The patient is not eligible or able to enrol in a clinical trial or continue participation in such trial.
4. There is a potential patient benefit to justify the potential risk of the treatment use, and the potential risk is not unreasonable in the context of the disease or condition to be treated.
5. The patient must meet any other medical criteria established by the medical experts responsible for the product or by the health authority in the country of request (as applicable).
6. Provision of the product will not interfere with the initiation, conduct, or completion of a Novartis clinical trial or overall development program.
7. Managed Access provision is allowed per local laws/regulations

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals